CLINICAL TRIAL: NCT04555512
Title: Efficacy of Prescription Methods for High-intensity Interval Training in Patients Enrolled in Outpatient Cardiac Rehabilitation
Brief Title: A Study to Compare the Effectiveness of Different High-intensity Interval Training Programs in Cardiac Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda R. Bonikowske, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-005923
Record Dates: First submitted 2020-09-03; First posted 2020-09-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-care interval-training group (Active Comparator): Subjects will complete a standard interval-training program that remains constant for the entire 12 weeks of cardiac rehabilitation.
  Interventions: Other: Constant High Intensity Interval Training (CON-HIIT)
- Progressive interval-training group (Experimental): Subjects will complete an interval-training program during which the number of intervals and the duration of each interval are changed across the 12-week cardiac rehabilitation program.
  Interventions: Other: Progressive High Intensity Interval Training (PRO-HIIT)

INTERVENTIONS:
Other: Progressive High Intensity Interval Training (PRO-HIIT) — Individual exercise training sessions, involving two weeks of moderate intensity continuous exercise and 10 weeks of interval exercise training. This protocol involves progression of training of 3 stages: 1) six high-intensity intervals (at an RPE of 15-18) of 1-min separated by five low-intensity intervals of 2-min; 2) three high-intensity intervals of 2-min separated by two low-intensity intervals of 4-min, and a further 2-min of low intensity following the last interval before cool-down; and 3) three high-intensity intervals of 3-min separated by two low-intensity intervals of 3-min, and a further 1-min of low intensity following last interval before cool-down.
  Arms: Progressive interval-training group
Other: Constant High Intensity Interval Training (CON-HIIT) — Individual exercise training sessions, involving two weeks of moderate intensity continuous exercise and 10 weeks of interval exercise training. This protocol involves a constant protocol of training, including six high-intensity intervals (at an RPE of 15-18) of 1-min separated by five low-intensity intervals of 2-min.
  Arms: Standard-care interval-training group

SUMMARY:
The purpose of the study is to examine the effect of two different high intensity interval training (HIIT) prescription approaches on improving fitness, heart function, and the ability of the body's muscles to receive oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older.
* English speaking.
* Able to provide consent.
* Has a qualifying indication for center-based cardiac rehabilitation that is non-surgical (i.e., Acute coronary syndrome, myocardial infarction, percutaneous coronary intervention, and stable angina).

Exclusion Criteria:

* Participants referred to cardiac rehabilitation following coronary artery bypass surgery, heart valve repair/replacement, heart transplant, or those with ventricular assist devices.
* Patients who are unable to engage in a regularly structured exercise training program as part of a clinically indicated center-based outpatient cardiac rehabilitation program are not eligible.
* Patients unable/unwilling to provide informed consent will not be enrolled.
* Patients identified as having a contraindication to high intensity exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorepiratory fitness | Pre and post study completion, approximately 12 weeks
  Measure as peak oxygen consumption (VO2 peak)

SECONDARY OUTCOMES:
Change in oxygen uptake response time | Weekly, over 12 weeks
  Measured as exponential time-constant of pulmonary oxygen uptake at exercise onset
Change in locomotor muscle oxygenation | Pre and post study completion, 12 weeks
  Measured as tissue oxygen saturation by near-infrared spectroscopy (NIRS)
Change in metaboreflex stimulation | Pre and post study completion, 12 weeks
  Measured as changes in blood pressure during recovery from exercise
Changes in mechanoreflex stimulation and sensitization | Pre and post study completion, 12 weeks
  Measured as changes in blood pressure during recovery from exercise
Change in cardiac function | Pre and post study completion, 12 weeks
  Measured as global longitudinal strain by echocardiography at rest and during sub-maximal exercise
Change in body composition | Pre and post study completion, 12 weeks
  Measured as fat mass by dual-energy x-ray absorptiometry
Change in blood pressure | Pre and post study completion, 12 weeks
  Measured as resting and mean 24-hr blood pressures by ambulatory blood pressure monitor
Change in blood lipids | Pre and post study completion, 12 weeks
  Measured as total-cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides
Change in physical activity | Pre and post study completion, 12 weeks
  Measured as minutes spent in moderate-vigorous physical activity, by accelerometer monitor

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Bonikowske, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials